CLINICAL TRIAL: NCT06971796
Title: Longitudinal Outcomes and Adherence of the Inspire System, EURO-STIM Registry
Brief Title: EURO-STIM Registry
Acronym: EURO-STIM
Status: Recruiting | Type: Observational
Sponsor: Inspire Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-004
Record Dates: First submitted 2025-04-07; First posted 2025-05-14 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea; Obstructive Sleep Apnea (OSA)
Keywords: Sleep Apnea; OSA; Inspire; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Device: Inspire UAS System — Participants will be implanted with the Inspire UAS System, which is a permanent, implantable therapy that consists of three implantable components: an IPG, a stimulation lead, and a sensing lead. In addition, the study subject receives a remote control to activate the therapy.

SUMMARY:
The registry is to measure longitudinal outcomes and adherence of the Inspire System. The goal of the registry is to capture the life cycle of the patient's use of the Inspire System through routine clinical care visits. There are no required interventions or testing.

ELIGIBILITY:
Inclusion Criteria:

Any patient implanted with or receiving an Inspire implant, who meets the following criteria, is eligible to participate in the registry:

1. Capable of giving informed consent, as required per institution
2. Willing to return for routine clinic visits as required for Inspire therapy management

Exclusion Criteria:

Any patient who meets any of the following criteria will not be eligible to participate in the registry:

1. Has a life expectancy of less than one year
2. Any reason the clinician deems patient is unfit for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously implanted or scheduled to be implanted with an Inspire System will be informed of the registry and given the option to participate by qualified Euro-Stim Registry staff. Up to 1,000 patients at up to 55 centers in multiple countries in the European Union and the United Kingdom will be included in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2035-04 (Estimated); Study Completion 2035-04 (Estimated)

PRIMARY OUTCOMES:
Apnea Hypopnea Index (AHI) | Total AHI, supine and non-supine AHI, documented as events/hour of sleep will be collected at baseline, prior to implant, and at follow-up visits, if available, as determined by clinical standard of care.
  The AHI, or number of apnea and hypopnea events per hour, is a measure of OSA severity.
Epworth Sleepiness Scale (ESS) | ESS will be collected at baseline and follow-up visits, if available, as determined by clinical standard of care.
  The ESS is a validated, self-report instrument that rates a subject's tendency to fall asleep in eight common daily situations13. The ESS has been validated primarily in OSA.

SECONDARY OUTCOMES:
DISE VOTE Classification | DISE VOTE Score will be collected, if available, at baseline.
  A Drug-Induced Sleep Endoscopy (DISE) is a diagnostic, standard of care procedure performed as part of the evaluation for airway surgeries (including implant of the Inspire System). The DISE is utilized to visualize the patient's airway obstruction.
Functional Outcomes of Sleep Questionnaire (FOSQ-30) | FOSQ-30 will be collected at baseline and follow-up visits, if available and only if already collected as part of routine clinical care.
  The FOSQ-30 is a validated, quality of life measurement that assesses the effect of a subject's daytime sleepiness on activities of ordinary living. It is commonly used in the clinical evaluation and management of OSA.
Patient Experience with Therapy (PET) | PET will be collected at follow-up visits after device activation, if available.
  The PET is a survey designed to collect information about patient's experience with the Inspire therapy.
Maintenance of Wakefulness Test (MWT) | Sleep latency is recorded in minutes and may be collected from a maintenance of wakefulness test performed at baseline and follow-up visits after device activation, if available.
  The maintenance of wakefulness test is used to measure a person's ability to stay awake during a defined period of time.
Therapy Use | Therapy use will be collected at follow-up visits after device activation, if available.
  Therapy use, reported as hours of use per week, is recorded during follow-up visits and will be collected from the Inspire physician programmer.
Adverse Events | The number of events (as well as the % of subjects in which the event occurred) will be reported at implant and at follow-up timepoints.
  Both serious and non-serious procedure-related and device/therapy related adverse events will be collected and reported.

CONTACTS AND LOCATIONS:
Locations (21):
- Austria (2):
  - Klinikum Klagenfurt, KABEG, Klagenfurt
  - Ordensklinikum Linz, Linz
- Universitair Ziekenhuis Antwerpen, Edegem, Belgium
- France (6):
  - Angers University Hospital Center, Angers
  - CHU Grenoble Alpes, La Tronche
  - Clinique de la Louviere, Lille
  - Hôpital d'Instruction des Armées Laveran, Marseille
  - Clinique Beausoleil, Montpellier
  - CHU Saint Etienne, Saint-Priest-en-Jarez
- Germany (6):
  - Asklepios Klinik Hamburg, Hamburg
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Klinik für HNO-Heilkunde/HNO-Schlaflabor, Lübeck
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg
  - Universitäts-HNO-Klinik Mannheim, Mannheim
  - Klinikum Rechts der Isar Technische Universität München, Munich
- Netherlands (2):
  - Sint Lucas Andreas Ziekenhus (OLVG), Amsterdam
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
- Kantonnspital Baselland-Liestal, Liestal, Switzerland
- United Kingdom (3):
  - Guy's & St Thomas' NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Manchester University NHS Trust, Manchester